CLINICAL TRIAL: NCT01318005
Title: The Effects of Dose and Formulation of Oral Contraceptives (OCs) on Breast-Cell Proliferation: Can the Chemopreventive Effects of OCs on Endometrial and Ovarian Cancer be Extended to Breast Cancer?
Brief Title: Oral Contraceptive (OC) Estrogen Dose and Breast Proliferation
Acronym: OCP2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Southern California (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: HS-10-00455
Record Dates: First submitted 2011-03-16; First posted 2011-03-18 (Estimated); Last update posted 2014-09-10 (Estimated); Status verified 2014-09

CONDITIONS: Oral Contraceptive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ortho-Novum® 1/35 (Active Comparator): Ortho-Novum® 1/35 is an oral contraceptive that contains more progestin.
  Interventions: Drug: Oral Contraceptive: Ortho-Novum® 1/35
- Ovcon® 35 (Active Comparator): Ovcon® 35 is an oral contraceptive that contains less progestin.
  Interventions: Drug: Oral Contraceptive: Ovcon® 35
- Microgestin Fe® 1/20 (Active Comparator): is an oral contraceptive that contains less estrogen.
  Interventions: Drug: Oral Contraceptive: Microgestin Fe® 1/20

INTERVENTIONS:
Drug: Oral Contraceptive: Ortho-Novum® 1/35 — Oral Contraceptive: Ortho-Novum® 1/35, pill, 2-3 mos, daily.
  Arms: Ortho-Novum® 1/35
Drug: Oral Contraceptive: Ovcon® 35 — Oral Contraceptive: Ovcon® 35, pill, 2-3 mos, daily.
  Arms: Ovcon® 35
Drug: Oral Contraceptive: Microgestin Fe® 1/20 — Oral Contraceptive: Microgestin Fe® 1/20, pill, 2-3 mos, daily.
  Arms: Microgestin Fe® 1/20

SUMMARY:
The purpose of this research study is to gain a better understanding of the changes that may occur in the breast when a woman uses an oral contraceptive (birth control pill). Some research indicates that women who use birth control pills with lower amounts of estrogen (a hormone in the birth control pill) may have lower breast cell growth than women who use birth control pills with a higher amount of estrogen; this research will examine that in detail. This research will also test whether the results found in HS-07-00269 can be confirmed.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-35
2. BMI <30 kg/m2
3. Premenopausal with regular cycles or currently taking an OC
4. Not currently or recently pregnant or nursing (within previous 6 months)
5. Non-smoker
6. No use of antibiotics within the prior 4 weeks
7. Competent to provide written informed consent (as judged by study team)
8. Willing to adhere to the OC regimen
9. Willingness to refrain from the use of aspirin or NSAIDS 10 days pior to the biopsy appointment and one week following the biopsy procedure
10. Willing and able to refrain from use of fish oils 10 days prior to the biopsy appointment and one week following the biopsy procedure

Exclusion Criteria:

1. Diabetes
2. Abnormal breast examination
3. Abnormal PT/INR and/or CBC with platelets test results (as determined by one of the study physicians)
4. History or current therapeutic or prophylactic use of anticoagulants
5. Known bleeding disorder or history of unexplained bleeding or bruising
6. History of breast cancer or previous diagnostic breast biopsy
7. Known allergy to local anesthetic

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 85 (Estimated)
Dates: Start 2011-01; Primary Completion 2015-06 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
To measure breast cell proliferation levels between the three oral contraceptive dose groups. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Heather MacDonald, M.D., Principal Investigator — University of Southern California
Locations (1):
- USC University Hospital, Los Angeles, California, United States